CLINICAL TRIAL: NCT05693753
Title: Coronally Advanced Flap With Xenogenic Collagen Matrix or Autogenous Connective Tissue Graft for the Treatment of Multiple Adjacent Gingival Recessions: a Randomized Controlled Trial
Brief Title: Xenogenic Collagen Matrix for the Treatment of Multiple Gingival Recessions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XCMTurin
Record Dates: First submitted 2023-01-11; First posted 2023-01-23 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Gingival Recession, Generalized
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xenogenic collagen matrix (XCM) (Experimental): Multiple coronally advanced flap technique (mCAF) with the use of a XCM
  Interventions: Device: Use of XCM for the treatment of MAGRs with mCAF technique
- Connective tissue graft (CTG) (Active Comparator): Multiple coronally advanced flap technique (mCAF) with the use of a CTG
  Interventions: Procedure: Treatment of MAGRs with CTG

INTERVENTIONS:
Device: Use of XCM for the treatment of MAGRs with mCAF technique — After local anaesthesia, mCAF technique will be performed. XCM will be adapted on the root surfaces and positioned at the level of the cemento-enamel junction.
  Arms: Xenogenic collagen matrix (XCM)
Procedure: Treatment of MAGRs with CTG — After local anaesthesia, mCAF technique will be performed. CTG will be adapted on the root surfaces and positioned at the level of the cemento-enamel junction.
  Arms: Connective tissue graft (CTG)

SUMMARY:
The primary aim of this study is to evaluate whether the use of a xenogenic collagen matrix (XCM) for the treatment of multiple adjacent gingival recessions (MAGRs) with a multiple coronally advanced flap technique (mCAF) achieves better results than the use of an autologous connective tissue graft (CTG) in terms of recession reduction (primary outcome) and other secondary root coverage outcomes (e.g. complete root coverage, mean root coverage). Moreover, this study aims to compare secondary clinical variables (e.g. keratinized tissue width (KTW) changes, probing pocket depth (PPD) changes, volumetric gain (VG), etc.), also with a digital approach, the patient-reported outcome measures (PROMs e.g. pain, swelling, bleeding). The hypothesis of this study is that at 6 months and 1 year follow-up the mCAF with XCM is not inferior to CTG in terms of recessions reduction and secondary clinical variables, and superior regarding to PROMs.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old and able to sign informed consent
* At least 2 adjacent teeth with RT1 and/or RT2 gingival recessions without interproximal exposure of the CEJ (interdental gingival recession), at least one with a depth of ≥2mm with indication for root coverage treatment
* A minimum of 4 adjacent teeth (including the ones to be treated) in the region of interest
* Available to attend study related procedures (including follow-up visits)

Exclusion Criteria:

* Systemic diseases/medications which could influence the outcome of the therapy (e.g., uncontrolled diabetes mellitus);
* Current smokers (self-reported, any type of smoking), users of chewing tobacco, and drug/alcohol abusers;
* Pregnant or nursing women;
* History of previous periodontal surgery (mucogingival or other) on the teeth to be included;
* Furcation involvement in the teeth to be included;
* Presence of severe tooth malposition, rotation or clinically significant extrusion in the teeth to be treated;
* Presence of fixed or removable prosthesis in the area to be treated

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2024-06-02 (Estimated); Study Completion 2024-12-02 (Estimated)

PRIMARY OUTCOMES:
Mean Recession Reduction (RecRed) | 6 months; 1 year
  Mean changes in mm in recession depth between baseline and 1-year

SECONDARY OUTCOMES:
Complete Root Coverage (CRC) | 6 months; 1 year
  Percentage of sites with complete root coverage after 1-year
Mean Root Coverage (MRC) | 6 months; 1 year
  Percentage of mean root coverage after 1-year
Keratinised tissue height (KTH) changes | 6 months; 1 year
  Linear changes in mm from the gingival margin to the mucogingival junction between baseline and 1-year
Post-operative morbidity (pain, swelling, discomfort) | 14 days
  Assessment of patient's pain, swelling and discomfort at 14 days after the procedure using visual analogue scale (VAS) ranging from 0 (no pain, swelling or discomfort) to 10 (maximum pain, swelling or discomfort) with a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- CIR Dental School, Turin, Italy

IPD SHARING:
Plan to Share IPD: Undecided